CLINICAL TRIAL: NCT07111338
Title: Telitacicept in the Treatment of Proliferative Glomerulonephritis With Monoclonal Immunoglobulin Deposits (PGNMID): A Prospective, Single-Arm Study
Brief Title: Telitacicept for PGNMID: A Single-Arm Study
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025R-0014; 2025SF047 (Other Grant/Funding Number: Peking University First Hospital)
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-02

CONDITIONS: Proliferative Glomerulonephritis With Monoclonal Immunoglobulin Deposits
Keywords: Telitacicept; PGNMID; proliferative glomerulonephritis; MGRS; BLyS/APRIL inhibitor
MeSH Terms: interventions — telitacicept

STUDY DESIGN:
Intervention Model Description: Single-group assignment: all eligible participants receive telitacicept 160 mg subcutaneously once weekly for 24 weeks without concurrent control or randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Telitacicept 160 mg Subcutaneous Once Weekly (Experimental): Participants receive telitacicept 160 mg by subcutaneous injection once weekly for 24 consecutive weeks. No placebo or active comparator is provided.
  Interventions: Drug: Telitacicept 160mg

INTERVENTIONS:
Drug: Telitacicept 160mg — Telitacicept (RC18) is a recombinant TACI-Fc fusion protein that simultaneously neutralizes B-lymphocyte stimulator (BLyS) and a proliferation-inducing ligand (APRIL), thereby inhibiting B-cell differentiation and plasma-cell survival. In this study, it is supplied as a sterile, preservative-free, lyophilized powder (160 mg/vial) that is reconstituted with 1 mL water for injection and administered subcutaneously into the abdomen or thigh at a fixed dose of 160 mg once weekly for 24 weeks. Each injection is performed by trained study personnel, and pre-filled backup syringes are available to ensure exact dosing. No dose escalation or tapering is planned; dose reductions or temporary discontinuation are allowed only for predefined safety criteria.

SUMMARY:
This single-center, prospective, single-arm study will evaluate the efficacy and safety of telitacicept in 10 adults with biopsy-proven proliferative glomerulonephritis with monoclonal immunoglobulin deposits (PGNMID).

Eligible participants (≥18 y, ≥1 g/day proteinuria, eGFR ≥20 mL/min/1.73 m²) will receive 160 mg telitacicept subcutaneously once weekly for 24 weeks after a 12-week run-in on maximally tolerated ACEi/ARB.

The primary endpoint is change in 24-hour urine protein from baseline to Week 24. Secondary endpoints include changes in eGFR, urine red-blood-cell count, and serum immunoglobulin/complement levels. Safety will be monitored throughout.

Recruitment is planned from May 2025 to May 2027 at Peking University First Hospital.

DETAILED DESCRIPTION:
Study Rationale Proliferative glomerulonephritis with monoclonal immunoglobulin deposits (PGNMID) is a rare but aggressive renal manifestation of monoclonal gammopathy of renal significance (MGRS). Conventional immunosuppression yields limited and inconsistent responses; no therapy is approved specifically for PGNMID. Pathogenic immunoglobulins are produced by dysregulated B-cell or plasma-cell clones. Telitacicept is a novel TACI-Fc fusion protein that simultaneously neutralizes B-lymphocyte stimulator (BLyS) and a proliferation-inducing ligand (APRIL), thereby suppressing both B-cell maturation and plasma-cell survival. This mechanism may interrupt the production of the monoclonal immunoglobulins that drive PGNMID.

Objectives Primary: To determine the change in 24-hour urine protein excretion from baseline to Week 24 after telitacicept therapy.

Secondary: (1) Change in estimated glomerular filtration rate (eGFR); (2) change in urinary red-blood-cell count; (3) change in serum IgG, IgA, IgM, C3, and C4; (4) safety and tolerability.

Study Design Single-center, open-label, investigator-initiated, prospective single-arm trial. Ten adults with biopsy-proven PGNMID will be enrolled. After a 12-week run-in on optimized ACE inhibitor or ARB therapy (to confirm persistent proteinuria ≥1 g/day), participants will receive telitacicept 160 mg subcutaneously once weekly for 24 consecutive weeks. Post-treatment follow-up continues to Week 28.

Population Inclusion: Age ≥18 y; renal biopsy consistent with PGNMID; 24-h proteinuria ≥1 g on two occasions ≥4 weeks apart despite maximal ACEi/ARB; eGFR ≥20 mL/min/1.73 m² (CKD-EPI); willingness to use effective contraception.

Exclusion: Malignant hematologic disorders (e.g., multiple myeloma); eGFR <20 or rapidly progressive GN; systemic immunosuppression within 3 months; active infection, hepatitis B/C, HIV; pregnancy/lactation; hypersensitivity to study drug.

Schedule of Assessments Screening (Weeks -12 to 0): medical history, physical exam, renal biopsy review, laboratory tests, informed consent.

Treatment period (Weeks 0-24): study drug administered at Weeks 0, 4, 8, 12, 16, 20, and 24. Laboratory panels, urinalysis, adverse-event (AE) assessment, and drug accountability will be performed at every visit.

Follow-up visit (Week 28): safety laboratory tests and AE collection. Endpoints & Statistical Plan Primary endpoint will be analyzed using a mixed-effect model for repeated measures (MMRM) with baseline proteinuria as covariate. Secondary continuous outcomes will be analyzed similarly. Descriptive statistics will summarize safety data. All participants who receive ≥1 dose will be included in safety analysis; modified intention-to-treat set will be used for efficacy. Missing data will be handled by multiple imputation. One-sided α = 0.05; no formal power calculation (exploratory study).

Safety Oversight An independent Data and Safety Monitoring Committee (DSMC) will review safety data every 3 months. Serious AEs will be reported to the institutional ethics committee and sponsor within 24 hours. A 24-hour emergency contact is provided to all participants.

Regulatory & Ethical Considerations The study is conducted in accordance with the Declaration of Helsinki and China's IIT guidelines. The Biomedical Research Ethics Committee of Peking University First Hospital approved the protocol (approval number：2025R-0014). Telitacicept is used off-label; this is explicitly detailed in the informed-consent form and hospital medical-affairs record.

Data Management Electronic case-report forms are maintained on a secure, password-protected server with daily back-ups. Only authorized study personnel have access. Participant identifiers are replaced by coded study IDs.

ELIGIBILITY:
Eligibility Criteria

**Inclusion Criteria**

1. Age ≥ 18 years
2. Renal biopsy consistent with proliferative glomerulonephritis with monoclonal immunoglobulin deposits (PGNMID) confirmed by central pathologic review
3. 24-hour urine protein ≥ 1 g on two occasions ≥ 4 weeks apart while receiving optimal renin-angiotensin system blockade (ACEi or ARB at maximal tolerated dose)
4. Estimated glomerular filtration rate (eGFR) ≥ 20 mL/min/1.73 m² calculated by CKD-EPI equation
5. Willing and able to provide written informed consent and comply with all study procedures

**Exclusion Criteria**

1. Rapidly progressive glomerulonephritis or crescentic disease (>50 % crescents)
2. Known malignant hematologic disorders (e.g., multiple myeloma, lymphoma)
3. Active malignancy (except adequately treated basal-cell carcinoma) within 5 years
4. Neutrophil count < 1.0 × 10⁹/L, hemoglobin < 80 g/L, or platelet count < 50 × 10⁹/L
5. ALT or AST > 2.5 × upper limit of normal (ULN) or total bilirubin > 1.5 × ULN
6. Chronic obstructive pulmonary disease (COPD) requiring systemic steroids or Stage III/IV heart failure (NYHA)
7. Systemic immunosuppressive or biologic therapy (e.g., cyclophosphamide, rituximab, bortezomib, lenalidomide, tacrolimus, mycophenolate, etc.) within 3 months prior to screening
8. Chronic or latent infection: active tuberculosis, HBV (HBsAg-positive or HBV-DNA-positive), HCV antibody-positive, or HIV-positive
9. Live vaccine within 4 weeks of screening
10. Known hypersensitivity to telitacicept or any excipients
11. Pregnancy, breastfeeding, or inadequate contraception (women of child-bearing potential and men not using highly effective contraception)
12. Any condition that, in the investigator's opinion, would compromise participant safety or interfere with study conduct

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-07-12 (Actual); Primary Completion 2027-05-29 (Estimated); Study Completion 2027-05-29 (Estimated)

PRIMARY OUTCOMES:
Change in 24-hour urine protein excretion from baseline to Week 24 | Baseline (Week 0) to Week 24
  Absolute change (g/24 h) in quantitative proteinuria from baseline (Week 0) to Week 24 after the first telitacicept dose, measured by 24-hour urine collection and averaged from two consecutive collections obtained within 7 days of the target visit.

SECONDARY OUTCOMES:
Change in estimated glomerular filtration rate (eGFR) from baseline to Week 24 | Baseline (Week 0) to Week 24
  Absolute change in eGFR (mL/min/1.73 m²) calculated with the CKD-EPI equation from baseline (Week 0) to Week 24.
Urinary Red-Blood-Cell Count | Time Frame: Baseline (Week 0) to Week 24
  Description: Absolute change in urinary RBC count (cells per high-power field) from baseline to Week 24, assessed in fresh morning urine by standardized microscopy.

OTHER OUTCOMES:
Serum Immunoglobulin Levels | Time Frame: Baseline (Week 0) to Week 24
  Description: Absolute change in serum IgG, IgA and IgM concentrations (g/L) from baseline to Week 24.
Serum Complement Levels | Time Frame: Baseline (Week 0) to Week 24
  Description: Absolute change in serum C3 and C4 concentrations (g/L) from baseline to Week 24.
Safety & Tolerability | Time Frame: Week 0 through Week 28
  Incidence and severity of treatment-emergent adverse events (CTCAE v5.0) during the 24-week treatment period plus 4-week follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Fude Zhou, MD, Study Director — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Renal Division, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Due to current regulations of the China Human Genetic Resources Administration (HGRAC), de-identified individual-level human genomic and clinical data cannot be transferred outside mainland China. While limited domestic sharing within China may be possible, international dissemination is restricted at this time.